CLINICAL TRIAL: NCT00193700
Title: Pharmacokinetic Evaluation of Testosterone Gel (1%) in Prepubertal Boys of Adolescent Age
Brief Title: Pharmacokinetic Evaluation of Testosterone Gel (1%)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: Unimed Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMD-01-080
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2006-12-25 (Estimated); Status verified 2006-11

CONDITIONS: Primary or Secondary Hypogonadism; Constitutional Delay in Growth and Puberty (CDGP)
Keywords: Hypogonadism
MeSH Terms: conditions — Hypogonadism

INTERVENTIONS:
Drug: Testosterone Gel (1%)

SUMMARY:
Measure and evaluate the level of testosterone in blood, and determine the safety and tolerability following daily applications of testosterone gel. Subjects who complete this trial may participate in the extension part (UMD-01-080E).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or secondary hypogonadism or constitutional delay in growth and puberty (CDGP)

Exclusion Criteria:

* Clinically significant uncontrolled medical condition or psychiatric disorder

Ages: 13 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (9):
- United States (9):
  - Site 208, Birmingham, Alabama
  - Site 203, Torrance, California
  - Site 204, Jacksonville, Florida
  - Site 201, Kansas City, Missouri
  - Site 206, Morristown, New Jersey
  - Site 207, Brooklyn, New York
  - Site 209, Cincinnati, Ohio
  - Site 202, Philadelphia, Pennsylvania
  - Site 205, Seattle, Washington